CLINICAL TRIAL: NCT02414464
Title: In-Office Tooth Bleaching for Young Patients Using a Hydrogen Peroxide-based Gel: a Randomized, Controlled, Clinical Trial
Brief Title: Tooth Bleaching for Young Patients Using a Hydrogen Peroxide-based Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBYP
Record Dates: First submitted 2014-12-09; First posted 2015-04-10 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Tooth Discoloration
Keywords: tooth bleaching; adolescent; clinical trial
MeSH Terms: conditions — Tooth Discoloration | interventions — Hydrogen Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 35% hydrogen peroxide (Experimental): Volunteers of this group will receive a gel with 35% hydrogen peroxide - Whiteness HP 35% for whitening treatment.
  Interventions: Other: 35% hydrogen peroxide
- 35% hydrogen peroxide with calcium (Experimental): Volunteers of this group will receive a gel with 35% hydrogen peroxide with calcium - Whiteness HP Blue Calcium 35% for whitening treatment.
  Interventions: Other: 35% hydrogen peroxide
- 20% hydrogen peroxide with calcium (Experimental): Volunteers of this group will receive a gel with 35% hydrogen peroxide with calcium - Whiteness HP Blue Calcium 20% for whitening treatment.
  Interventions: Other: 20% hydrogen peroxide

INTERVENTIONS:
Other: 35% hydrogen peroxide — Prophylaxis was performed with a jet of sodium bicarbonate to remove extrinsic pigments and plaque.
  Each patient underwent two bleaching sessions. A lip retractor (Arc Flex, FGM®) was placed. Cotton roles or gauze compresses were used to achieve relative isolation. A dental dam (Top Dam, FGM®) was placed over the free marginal gingival tissue and the inter-tooth papillae of teeth 14 to 24 in each session. The Whiteness HP 35% gel was applied to the vestibular faces of these teeth.
  In the present study, the Whiteness HP 35% gel was applied without an external auxiliary source. As this is not a self-catalyzed system, the gel was removed after each 15-minute application and reapplied two more times, totaling 45 minutes of contact with the teeth.
  Other Names: Whiteness HP 35%
  Arms: 35% hydrogen peroxide
Other: 35% hydrogen peroxide — Prophylaxis was performed with a jet of sodium bicarbonate to remove extrinsic pigments and plaque.
  Each patient underwent two bleaching sessions. A lip retractor (Arc Flex, FGM®) was placed. Cotton roles or gauze compresses were used to achieve relative isolation. A dental dam (Top Dam, FGM®) was placed over the free marginal gingival tissue and the inter-tooth papillae of teeth 14 to 24 in each session. The Whiteness HP Blue Calcium 35% gel was applied to the vestibular faces of these teeth for 40 minutes in each session.
  Other Names: Whiteness HP Blue Calcium 35%
  Arms: 35% hydrogen peroxide with calcium
Other: 20% hydrogen peroxide — Prophylaxis was performed with a jet of sodium bicarbonate to remove extrinsic pigments and plaque.
  Each patient underwent two bleaching sessions. A lip retractor (Arc Flex, FGM®) was placed. Cotton roles or gauze compresses were used to achieve relative isolation. A dental dam (Top Dam, FGM®) was placed over the free marginal gingival tissue and the inter-tooth papillae of teeth 14 to 24 in each session. The Whiteness HP Blue Calcium 20% gel was applied to the vestibular faces of these teeth 50 minutes in each session.
  Other Names: Whiteness HP Blue Calcium 20%
  Arms: 20% hydrogen peroxide with calcium

SUMMARY:
The aim of the present study was to evaluate colorimetric changes and tooth sensitivity in young patients submitted to tooth bleaching with 20% and 35% hydrogen peroxide.

DETAILED DESCRIPTION:
A randomized, controlled, clinical trial was conducted with 53 patients aged 11 to 24 years who were allocated to groups based on the use of the following commercial products: Whiteness HP - FGM® (35% hydrogen peroxide); Whiteness HP Blue Calcium - FGM® (35% hydrogen peroxide); and Whiteness HP Blue Calcium - FGM® (20% hydrogen peroxide).

After the bleaching procedure, the visual analog scale was used to measure tooth sensitivity and the classic Vita® scale was used to determine changes in tooth color.

Statistical analysis involved the Friedman, Kruskal-Wallis and Student-Newman-Keuls tests, with p-value ≤ 0.05 or ≤ 0.0001 considered indicative of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 11 to 24 years with a diagnosis of tooth discoloration and a signed statement of informed consent.

Exclusion Criteria:

* Individuals with dentofacial anomalies, those without the permanent dentition complete to the second molars, those in orthodontic or orthopedic treatment of the jaws, those who took medications that could alter tooth color and those who had previously been submitted to tooth bleaching

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Discoloration | Change of teeth color after 48 hours, after 6 months, after 12 months, after 18 months
  the initial tooth color was determined with the aid of the classic Vita® scale. Tooth color was recorded 48 hours after each session to determine the difference in tone before and after the procedures.
  It will be carried out in all groups at the following times: pre-treatment period, 48 hours following each session, after six months, after 12 months, after 18 months.

SECONDARY OUTCOMES:
Dental sensitivity | Sensivity alteration up to 48 hours after the procedure
  The visual analog scale was used for the subjective measure of sensitivity during and after the procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Bussadori, Doctor, Study Director — University of Nove de Julho